CLINICAL TRIAL: NCT01226992
Title: Phase II/III Randomized Controlled Trial of Oral Vancomycin Followed by Fecal Transplantation Versus Tapering Oral Vancomycin for Recurrent Clostridium Difficile Infection (CDI)
Brief Title: Oral Vancomycin Followed by Fecal Transplant Versus Tapering Oral Vancomycin
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unavailable study resources
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UHN # 08-0440; 9424-U0288/2-25C 124081 (Other: Health Canada)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-10

CONDITIONS: Recurrent Clostridium Difficile Infection; Laboratory Confirmed Clostridium Difficile Infection
Keywords: Clostridium difficile; Fecal Transplant; Recurrent Diarrhea; Abdominal distension/bloating; Fever
MeSH Terms: conditions — Clostridium Infections; Diarrhea; Fever | interventions — Vancomycin; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal Transplant (Experimental): 2 weeks of oral vancomycin pre-treatment followed by single dose fecal transplant administered by rectal enema. Fecal transplant (slurry) consists of 50 grams healthy donor stool blended in 500ml of Normal Saline.
  Interventions: Biological: Fecal Transplant
- Oral Vancomycin Taper (Active Comparator): 2 weeks of oral vancomycin pre-treatment followed by 6-week taper of oral vancomycin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Oral Vancomycin:
  Dose: 125 mg po qid x 2 weeks then 125 mg po bid x 1 week then 125 mg po od x 1 week then 125 mg po q every other day x 1 week then 125 mg po q every third day x 1 week then discontinue Route: oral
  Arms: Oral Vancomycin Taper
Biological: Fecal Transplant — Fecal slurry 50 grams stool in 500ml normal saline
  Arms: Fecal Transplant

SUMMARY:
Recurrent CDI is a growing problem with few treatment options that provide lasting effect. Fecal transplantation has been shown in several case series to be successful in controlling recurrent CDI. The current study is a non-blinded, randomized controlled trial comparing fecal transplantation with a 6 week taper of oral vancomycin for the treatment of refractory CDI. Approximately 146 patients will be enrolled over one year. Participants in the study will be followed for 120 days, and will be given the opportunity to cross over to the alternative intervention arm if a relapse in symptoms occurs. The primary outcome measure will be recurrence of toxin-confirmed CDI within 120 days of starting the intervention. Secondary outcomes include: early recurrence of symptoms within 14 days, relapse within 120 days (same strain of C. difficile), attributable mortality, hospitalization and serious adverse events.

DETAILED DESCRIPTION:
The proposed trial is a single-centre, phase II/III, open, parallel-group, randomized controlled trial. To have an evaluable population of 114 participants and assuming a 20% loss to follow-up, approximately 146 patients will be randomized in a 1:1 ratio to receive either approximately 2 weeks of oral vancomycin followed by a single fecal transplant via enema (hereon referred to as the "fecal transplant arm") or a 6-week taper of oral vancomycin (hereon referred to as the "vancomycin taper arm"). The 2 weeks of vancomycin pre-treatment in the fecal transplant arm will allow for a fecal transplant donor to be screened for potentially transmissible infectious diseases (clinically and through blood and stool tests), in order to ensure appropriateness and safety of donation.

If patients fail treatment during the follow-up period of 120 days, they will be offered the opportunity to cross over to the alternate treatment arm. Those who cross over will be followed for an additional 120 days from the second intervention.

Participants will be assessed clinically for recurrence in CDI symptoms and adverse events at the following time points after the intervention: 4 days, 7 days, 3 weeks, 6 weeks, 12 weeks and 16 weeks. All recurrences of CDI symptoms will be investigated with C. difficile laboratory testing to confirm the etiology of these symptoms.

Analysis will be intention to treat. An interim analysis may take place after completion of follow-up of 30 patients. This interim analysis is meant to establish the safety and feasibility of the study, not measure efficacy. Although there were no formal sample size calculations to assess safety of the procedure, with a sample size of 70 participants, an adverse event rate, for example of 2.5%, can be detected with a probability of 0.83 for the fecal transplantation group.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory or pathology-confirmed diagnosis of recurrent C. difficile infection (CDI) with symptoms within the previous 60 days. Recurrent CDI is defined as:

  * >/=2 episodes of CDI. Eligible patients must have had at least one treatment course with oral vancomycin (minimum 10 days of 500 mg total daily oral vancomycin).

Symptoms of CDI include:

* Diarrhea (see below) OR
* Abdominal pain AND abdominal distension/bloating AND fever, systemic illness with no other reason for these symptoms

Diarrhea will be self-reported and is defined as:

* at least 6 watery feces in 36 hours OR
* 3 unformed feces in 24 hours for minimum 2 days OR
* 8 unformed feces over 48 hours

  * Age 18 years or older
  * Signed informed consent
  * Able to travel to clinic for follow-up visit and/or adhere to study procedures
  * Agrees to abstain from taking probiotic supplementations for medicinal reasons for the duration of the study and follow-up period. To clarify, dietary intake is acceptable (e.g. non-supplemented yogurt).

Exclusion Criteria:

* Planned participation in another clinical trial
* Patients with conditions such as neutropenia, graft versus host disease or severe immunocompromise, in whom enemas are contraindicated
* More than one episode of CDI that has been severe or rapid in onset, resulting in:

  * intensive care unit admission
  * Evidence of active, severe colitis (ie. ongoing diarrhea not responsive to oral vancomycin; hemorrhagic colitis) such that an enema is contraindicated (note that such patients may be eligible once their colitis is under control)
  * Unable to tolerate fecal transplantation procedure for any other reason
  * Hypersensitivity or intolerance to oral vancomycin
  * Patients with underlying chronic gastrointestinal diseases that cause diarrhea, such as:
  * Inflammatory bowel disease
  * Short gut syndrome
  * Severe motility disorders
  * Severe diverticular disease
  * Other chronic diarrhea NYD
  * Unable to record frequency of bowel movements
  * Receiving an investigational medication
  * Planned therapy in the next 120 days that may cause diarrhea (example: chemotherapy)
  * Planned surgery requiring perioperative antibiotics within 120 days
  * Pregnancy
  * Requires the regular use of medications that affect bowel motility before onset of CDI (example: metoclopramide, narcotics, loperamide)
  * Serious bleeding disorder, anticoagulant use that cannot be stopped temporarily for procedure (in consultation with prescribing physician) or serious platelet disorder (platelet counts below 50).
  * Any condition that, in the opinion of the investigator, would pose a health risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
A Randomized Controlled Trial of Oral Vancomycin Followed by Fecal Transplantation versus Tapering Oral Vancomycin Treatment for Recurrent Clostridium difficile Infection. | 3 years
  To assess the number of patients with recurrence of laboratory-confirmed CDI in the 120 days following completion of intervention with either oral vancomycin followed by fecal transplantation or a 6-week taper of oral vancomycin.

SECONDARY OUTCOMES:
A Randomized Controlled Trial of Oral Vancomycin Followed by Fecal Transplantation versus Tapering Oral Vancomycin Treatment for Recurrent Clostridium difficile Infection. | 3 years
  To evaluate the safety profile of fecal transplantation.
  To characterize other outcomes of patients treated with fecal transplantation and oral vancomycin, as determined by the following:
  i. Early (within 14 days of treatment completion) and late (within 120 days of treatment) recurrence of symptoms compatible with CDI; ii. Days with diarrhea in the 120 days post-treatment; iii. CDI requiring hospital admission in the 120 days after treatment onset; iv. All-cause and CDI-attributable mortality; v. Recurrence of CDI in the 120 days after crossover to the alternate treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Susy Hota, MD FRCPC, Principal Investigator — Infectious Disease, Infection Prevention and Control, Epidemiologist; Susan Poutanen, MD MPH FRCPC, Study Director — Infectious Disease, Microbiologist
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hota SS, Sales V, Tomlinson G, Salpeter MJ, McGeer A, Coburn B, Guttman DS, Low DE, Poutanen SM. Oral Vancomycin Followed by Fecal Transplantation Versus Tapering Oral Vancomycin Treatment for Recurrent Clostridium difficile Infection: An Open-Label, Randomized Controlled Trial. Clin Infect Dis. 2017 Feb 1;64(3):265-271. doi: 10.1093/cid/ciw731. Epub 2016 Nov 9. PMID 28011612